#### Official Title:

Fecal Microbiota Transplantation in the Treatment of
Inflammatory Bowel Disease: the Role of Selection of the Bai
Nationality as Donor Source in Terms of Treatment Efficacy
and Mechanisms

Date: September 8, 2024

#### **Study Protocol**

#### 1. Background

Inflammatory bowel disease (IBD) is a chronic, recurrent, non-specific intestinal disease, including ulcerative colitis (UC) and Crohn's disease (CD). Although biological therapy significantly improved the effect of the treatment of ulcerative colitis, but nearly two-thirds of the patient's response to drug treatment. Therefore, new treatments targeting the underlying pathophysiology of UC are critical. Given that alterations in the gut microbiome are strongly associated with disease activity in IBD, many studies have proposed microbiotoy-based therapies, in particular, Fecal microbiota transplantation (FMT) in the treatment of UC. Donor-to-donor variation in treatment with fecal microbiota transplantation may alter treatment efficacy. Therefore, screening high-quality donors can improve efficacy and minimize the risk of adverse effects.

Ulcerative colitis with the changes in the gut microbiota and biodiversity decrease and the change of the relative abundance of advantage bacterium group, a significant reduction in UC patients with intestinal flora diversity, at the species level, thick wall bacteria door bacteria (e.g., clostridium tender) ratio decreases, actinomyces door, the door deformation bacteria such as e. coli), enterobacteriaceae, Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: the Role of Selection of the Bai Nationality as Donor Source in Terms of Treatment Efficacy and Mechanisms September 8, 2024

streptococcus, bacteroides ratio increased. A previous study by team of the investigators found that there were ethnic and regional differences in the incidence of IBD in Yunnan Province, and the incidence of Dai, Bai and Miao was lower than that of Han. Then the related factors were analyzed, among which, the ethnic characteristic diet of Yunnan ethnic minorities can improve the diversity of intestinal flora and viruses, increase the content of probiotics, and is a protective factor for the low incidence of UC.Based on this, donor-to-donor variation in the treatment of fecal microbiota transplantation may alter the therapeutic effect. Therefore, screening high-quality donors can improve efficacy and minimize the risk of adverse effects. Based on this, the investigators asked scientific questions: FMT in the treatment of IBD: the Bai nationality of Yunnan province may be a high quality donor. Our study is aims to FMT in the treatment of IBD, the role of selection of the Bai nationality as donor source in terms of treatment efficacy and mechanisms.

#### 2. Objectives

#### 2.1 Primary Outcome

The primary outcome is a composite of steroid-free clinical remission together with endoscopic remission or response at week12, defined as defined as a total Mayo score of ≤2 points with no individual sub-score >1 point, and at least a 1 point reduction from baseline in the Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: the Role of Selection of the Bai Nationality as Donor Source in Terms of Treatment Efficacy and Mechanisms September 8, 2024

endoscopy sub-score.

#### 2.2 Secondary Outcome

i.Steroid-free clinical remission (defined as combined Mayo sub-scores of 1 or less for rectal bleeding plus stool frequency)

ii.Steroid-free clinical response (defined as either a decrease of 3 points or more on the Mayo score, a 50% or greater reduction from baseline in combined rectal bleeding plus stool frequency Mayo sub-scores, or both)

iii.Steroid-free endoscopic response (defined as a Mayo endoscopy sub-score of 1 or less, with a reduction of at least 1 point from baseline) iv.Changes in microbial composition (including bacteriome, virome and fungome), function and metabolite at weeks 0, 1, 8, 12

v.Change in microbiome of stool (including bacteriome, virome and fungome) at weeks 0, 1, 8, 12 and duration of change before reverting to baseline

vi.Difference in microbiome (including bacteriome, virome and fungome) compared between subjects in different treatment arm vii.Proportion of microbiome (including bacteriome, virome and fungome) derived from recipient, donor or both in subjects who received FMT

viii.Difference in microbiome (including bacteriome, virome and Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: the Role of Selection of the Bai Nationality as Donor Source in Terms of Treatment Efficacy and Mechanisms

September 8, 2024

fungome) compared between subjects who have weight loss and those do not have weight loss

ix.Microbial factors (including bacteriome, virome and fungome) that are associated with percentage of body weight loss

x.Trans-kingdom correlation of microbial engraftment after FMT between bacteriome, virome and fungome

| Groups (30 Patients/Group) | Samples | Before FMT<br>Day | Follow Up<br>(Week) | Follow Up<br>(Week) | Follow Up<br>(Week) |
|---|---|---|---|---|---|
| (30 Patients/Group) | | Baseline(0) | 1 | 8 | 12 |
| Fresh<br>(the Bai nationality<br>Donor) | Stool<br>and Urine<br>Blood<br>and Biopsies | √<br>√ | √<br>√ | √ | √<br>√ |
| Fresh | Stool<br>and Urine | $\checkmark$ | J | ✓ | √ |
| (the Han nationality<br>Donor) | Blood and Biopsies | √ | √ | | $\checkmark$ |

#### 3. Design

#### 3.1 FMT:

Fresh fecal bacterial solution was obtained through a fecal bacterial transplantation isolation system (FMT-6A-50/12-AS, Nanjing), which was directly infused into the ileocecal region through colonoscopy tube (100 mL each time) within 30 minutes. A total of 3 transplantations were performed on the 1st, 3rd and 5th day of admission, respectively. The fresh bacterial solution administered during the 3 FMT sessions was obtained from feces with a total weight of 100 g.

#### 3.2 Mayo score

Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: the Role of Selection of the Bai Nationality as Donor Source in Terms of Treatment Efficacy and Mechanisms September 8,2024

| Item | Score | Evaluation |
|---|---|---|
| 1. Stool frequency | 0 | Normal number of stools |
| | 1 | 1-2 more than normal |
| | 2 | 3-4 more than normal |
| | 3 | ≥ 5 more than normal |
| 2. Rectal bleeding | 0 | No blood seen |
| | 1 | Streaks of blood with stool in in less |
| | | than half of the cases |
| | 2 | Obvious blood with stools in most of |
| | | the time |
| | 3 | Blood alone passed |
| 4. Endoscopic findings | 0 | Normal mucosa or inactive disease |
| | 1 | Mild activity (erythema, decreased |
| | | vascular pattern, mild friability) |
| | 2 | Moderate activity (marked |
| | | erythema, lack of vascular pattern, |
| | | friability, erosions) |
| | 3 | Severe activity (spontaneous |
| | | bleeding, large ulcerations) |
| 5. Physician's global | 0 | Normal |
| assessment | 1 | Mild disease |

| 2 | Moderate disease |
|---|------------------|
| 3 | Severe disease |

#### 3.3 The clinical laboratory

Blood sampling for routine blood test, blood biochemistry, c-reactive protein (CRP) and blood sedimentation (ESR) detection.

#### 3.4 Histologic assessment

Colonic biopsy will adopt a colonoscopy histologic evaluation.

#### 6. Methods

Single-center randomized trial

6.1 Sample processing methods

The procedures of sample collections and subpackaging are as follows

- ① Study blood : Red heparin tube 5mL+Purple heparin tube 4mL.Centrifuge at centrifugal force of 2500 rpm and temperature of 4  $^{\circ}$ C for 15min, and finally subpackage in 2ml cryogenic vials.
- ②Study stool: The feces of patients are collected and packed into 2ml cryogenic vials.
- ③Study urine: Urine from patients was collected and then packed into a 15ml saliva tube.
- ④ Study biopsies: Two of the most severe rectal (10cm local anus) lesions are selected and placed in 2ml cryogenic vials.

#### 6.2 Fecal Calprotectin

Fecal calprotectin concentrations will be assessed in batches when Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: the Role of Selection of the Bai Nationality as Donor Source in Terms of Treatment Efficacy and Mechanisms

September 8, 2024

sufficient fecal samples have been collected for QUANTA Lite calprotectin ELISA assays. This is an enzyme-linked immunosorbent assay (ELISA) system that is based on colorimetric detection of polyclonal antibodies to calprotectin. The enzyme-linked immunosorbent assay ranged from 10 to 1800 mg/g. The required sample volume ranged from 50 to 150ml, and the test sensitivity was less than 10mg/g. The treatment arm of the subject will be analyzed in a blinded manner.

#### 6.3 Microbiological Analysis

#### (1) Extraction of nucleic acids

DNA was isolated from the study samples using Maxwell® RSC PureFood GMO and Authentication Kit according to protocol. Fecal pellets were first added to CTAB buffer and vortex and heated for 5 min. Proteinase K and RNase A were added to the samples and incubated at  $70\,^{\circ}\text{C}$ . After centrifugal, collecting supernatant, transferred to Maxwell ® RSC instrument.

#### ② Microbial and metabolomic analysis

The collected specimens will undergo laboratory microbiological analysis, including bacterial, viral, and fungal components of the human microbiome. Qiagen QIAamp®DNA Mini Kit, Qiagen QIAamp DNA Stool Mini Kit, Mobio UltraClean®Tissue & Cells DNA Isolation were used Kit, Maxwell®RSC PureFood GMO, and Authentication Kit perform different DNA enrichment and extraction methods for bacteria, viruses, and fungi. Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: the Role of

Subsequent metagenomic sequencing was performed with the use of a Novoseq 6000 (2x300bp double-ended) system. Bacteria, fungi, and viruses were analyzed by methplan2, UNITE2-Bowtie2, and Kraken2, respectively. DESeq, Random Forest, and LEfSe linear discriminant analysis will be used to compare the differences in microbiome, metabolome, and metatranscriptome configurations between treatment groups, donors, and specimens at different time points. DESeq and Random Forest are executed in R via the DESeq and randomForest packages, respectively. Lefse analysis will be hutten hall lab galaxy server (http://huttenhower.sph.harvard.edu/y/). A DB-RDA analysis will be performed in R to describe the influence of other clinical factors on polysomy.

#### 6.4 Studies in Animals

Animal studies may be performed using collected biological samples. For example, fecal samples collected from FMT donors and recipients can be gavaged into animal models to study the effects of the microbiota.

| 7. Clinical study approval document issued by the Ethics Committee of |
|-----------------------------------------------------------------------|
| the First Affiliated Hospital of Kunming Medical University |

### Clinical study approval document issued by the Ethics Committee of the First Affiliated Hospital of Kunming Medical University

(2023) Lun L No. 127

| | (2023) Edil E NO. 121 |
|---|---|
| project<br>name | Mechanism and clinical study of fecal bacteria transplantation for inflammatory bowel disease |
| Application<br>Authority<br>(person) | The First Affiliated Hospital of Kunming Medical University |
| Undertake<br>the<br>department | department of Principal gastroenterol investigato ogy According to should rayZhang of chief physician al ranks and title s |
| Source of<br>research<br>funds | ■ Government mouth Foundation Kou Company□ international cooperationD. Others (please indicate) |
| Send review<br>documents | 1 Study protocol (Version No:1.0. Date: June 7,2023) 2 Informed Consent Form (Version 1.0, dated 07 June 2023) 3 Case Report Form (Version No.1.0, dated 07 June 2023) 4 CV of principal investigator and copy of GCP training certificate |
| Ethical | □ Conference Review |
| revie | ■ Quick Review |
| w | |
| metho | |
| ds | |
| juror<br>Review | Du Qinglin and Zhang Ling |
| comments | Agreed to proceed at this center, |
| from the | |
| Ethics | |
| Committe | |
| е | |
| | lities, personnel composition, operating procedures and records of ICH-CCP and relevant laws and regulations of China. |
| 1. The clinica of the ethic 2The study sho Committee and 3. From the da 12 months progress), expiration 4. During the consent for application the amendme 5. In case of | I test shall be implemented within 1 year from the date of approval s Committee, but not implemented during the fishing period. Several pieces of this review are be abolished. Utility the principles of CFD / CP and CP the of consent to the study, conduct regular follow-up visits every (the review compliance may change according to the actual please submit to the Ethics Committee one month before the of the regular review ( study. Any modifications to the study protocol and the informed rm. Please submit the relevant information in the amendment a form and the "submission document elimination form", and submit ent to the Ethics Committee before implementation. a serious adverse event or unexpected adverse event affecting the it ratio of the study, the Ethics Committee shall be reported to |
| the CDA in writing, using the CHDA (Serious Adverse Event Report Form or the Ethics Committee (Serious AE / Unanticipated AE Report Form or other relevant report forms, but the foreign language report requires a Chinese abstract, and the Ethics Committee has the right to make new decisions on its evaluation. | |
| | r violate the program should be timely not do or violate the program report |
| | termination of the study shall submit the |
| Termination Report Form of the study protocol in time. | |
| 8. Submit after the completion of selenium research ("Study Conclusion Report Form". | |
| | en report on important decisions of some thick conmittees. |
| | Chairman Sign e of Chairman: good i es Committee he 10th Affiliated Tosp (man) Medical University (man) |
| 1 | |
| Address: No | In 2 0 2 3, August 2 4<br>295, Xichang Road, Kunming, Yunnan province: 650032 Tel: 087i- |

#### 8. Statistical Analysis Plan

Continuous variables to mean (SD), said with a paired t test to compare the difference between the two groups. Classification variables will be compared using chi-square test or Fisher's exact test. The modified intention-to-treat analysis included all subjects receiving at least one FMT treatment. Patients who required treatment escalation, violated the study protocol, failed to discontinue corticosteroids at week 8, or discontinued the study for any reason were considered to have treatment failure. Each protocol analysis will include all patients who completed the 8-week masked study treatment course without protocol violation. Missing data will be used before the last observation to the method of calculation, so the missing values will be the last one is not the missing value replacement. A two-sided p value of less than 5% was considered to indicate statistical significance. Security will use descriptive statistical methods to collect data. All statistical tests were performed using SPSS Statistics version 20 (IBM Corporation, Armonk, NY).

| 9. Clinical study approval document issued by the Ethics Committee of |
|-----------------------------------------------------------------------|
| the First Affiliated Hospital of Kunming Medical University |

## The First Affiliated Hospital of Kunming Medical University

## Informed consent form for microflora transplantation (FMT / miniFMT)

surname and administrative Bed number: bed Hospitalization Number: Date: personal name: or technical offices:

| <b>D</b> : | 1.4. | .1 4 4 4 | | 1 |
|------------|---------------|-------------|------------|-----------|
| Disease | conditions an | a treatment | r recommen | idations: |

| | informationse: | | | | | |
|---|---|---|---|---|---|---|
| _ | | | | | Pregnancy history | v: 🗆 with 🗆 |
| Numbe | r of previo | ous FMT t | reatments: | (times), with | or without adverse | effects: 🗆 |
| □ not h | ave | | | | | |
| FMT Pro | e-treatme | nt examin | ation: | | | |
| ALT | U /L ; | AST | U /L ; | CRPmg/L; | ESRmm | ; |
| EB -DNA | ACo <sub>j</sub> | py/ml;HC | MV-DNA | copy /ml; | | |
| Stool ro | outine + o | ccult bloo | d: []; | | | |
| HbsAg [ | ]; An | ti -HBs [ | ]; HbeAg [ | ]; Anti -Hbe [ | ]; Anti -Hbc [ | ]; |
| Anti-HC | V []; Anti-H | IV 1 / 2 []; S | Syphilis: []; Other | rs: [] | | |
| 2. Trea | tment reco | ommenda <sup>s</sup> | tions | | | |
| I have ob | otained the | e following | g explanations: | microflora tran | splantation includes | fecal |
| bacteria trans | splantatio | n (FMT) ar | id formula mic | roflora transplaı | ntation (miniFMT or | SMT), |
| the indication | ns for micr | oflora trai | nsplantation, fo | oreign and dom | estic applications ar | nd |
| research stat | us, the ber | nefits for t | he diagnosis a | nd treatment of | diseases, the chanc | es of |
| surgical (or re | egimen) tr | eatment s | uccess, | | | |
| Including: the | e benefits | of function | nal intestinal flo | ora reconstruction | on, the recent impro | vement o |
| cure probabi | lity of the | disease, th | ie long-term ev | olution of the c | lisease, different dis | eases and |
| no | | | | | | |
| | , | | , | | ds of success during | • |
| treatment, ar | _ | | - | - | r has told me that I | |
| | | | | | e condition, faecal b | acteria |
| transplant | ation (FM | T / miniFM | IT) treatment o | an be performe | d. | |

## Our hospital has clearly informed the patient (close relatives / guardians) of the following contents:

(1) Although doctors have tried to eliminate possible risks, there may still be the risk of disease infection, "window period" problems that cannot be detected, wrong test results, and unpredictable risks; formula flora transplantation may also have unpredictable risks.

- (2) Possible main risks and complications in the process of microflora transplantation and related diagnosis and treatment, including failure of operation, perforation, bleeding, abdominal infection, etc. In case of occurrence, agree to the doctor to give the corresponding diagnosis and treatment disposal.
- (3) After the microflora transplant, my disease may be cured, partially effective, recurrent, or recurrent. Repeat implementation of microflora transplantation therapy may be required. I can choose to abandon this treatment strategy at any stage.
- (4) For the diagnosis and treatment needs of the condition, the members of the diagnosis and treatment team can implement relevant alternative diagnosis and treatment measures.

| Patients (close relatives / g | guardians) | include the | following | contents: |
|---|---|---|---|---|
|---|---|---|---|---|

| (1) I agree to and authorize it | (Physician signature) And its diagnosis and |
|---|---|
| treatment team to implement the fol | owing possible options: via colonoscopy, on |

Department of Gastroenterology, the First Affiliated Hospital of Kunming Medical University2Informed consent form for microflora transplantation (FMT / miniFMT)

# The First Affiliated Hospital of Kunming Medical University

## Informed consent form for microflora transplantation (FMT / miniFMT)

surname and administrative Bed number: bed Hospitalization Number: Date: personal name: or technical offices:

Gastrointestinal endoscopy, middle gastrointestinal endoscopy, gastric tube, nasojejunal tube, enema, oral capsule containing intestinal bacterial fluid, fistula tube, rectal graft tube (TET) (the involved endoscopy and anesthesia informed consent were signed separately).

- (2) The type of transplanted bacteria I received was: □ fresh fecal bacteria □ frozen fecal bacteria □ formula bacteria.
- (3) For faecal bacteria transplantation, I agree that the source of faecal bacteria is: 

  relatives 

  friends 

  Other healthy people, as suggested by the doctor. For formula flora transplantation, I knew that the group selection was determined by the doctor.
- (4) I agree that the hospital will preserve and use my fecal bacteria, body fluids and tissue specimens for teaching and medical research without involving personal identifiable information and privacy.
- (5) Each doctor and patient shall hold one copy of this informed consent. I have been told that the property right of this document belongs to the institute and shall not be issued and distributed without permission.
- (6) After full notification, I have read or passed my relatives have read and explained the above content, and I hereby sign the informed consent form.

#### Patients (close relatives / guardians) carefully promise that:

| Patient (close relative / guardi | an) signatı | ure: Relations | ship: Time: | year | moon |
|---|---|---|---|---|---|
| sun | | | | | |
| Doctor Signature: Time: | year | moon | sun | | |

| Department of Gastroenterology, the First Affiliated Hospital of Kunming Medical University <sup>2</sup> Informed consent form for microflora transplantation (FMT / miniFMT) |
|---|

# The First Affiliated Hospital of Kunming Medical University Informed consent form for microflora transplantation (FMT / miniFMT)

surname and administrative Bed number: bed Hospitalization Number: Date: personal name: or technical offices:

#### Commitment content

(I) My name is XXX, and I have understood the process and related risks of fecal transplantation. I strongly require fecal transplantation treatment, and I am willing to take all the risks.

(Family member) I am XXX from XXX. I have understood the process and related risks of fecal transplantation, so I strongly demand the treatment of fecal transplantation, and I am willing to take all the risks. Department of Gastroenterology, the First Affiliated Hospital of Kunming Medical University2Informed consent form for microflora transplantation (FMT / miniFMT)